CLINICAL TRIAL: NCT02475096
Title: Internet-delivered Cognitive Behavior Therapy for Children With Pain-predominant Functional Gastrointestinal Disorders - an Open Pilot Study
Brief Title: Internet-delivered CBT for Children With Functional Gastrointestinal Disorders - an Open Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Ola Olen, PhD MD, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pilot child ICBT FGID
Record Dates: First submitted 2015-06-15; First posted 2015-06-18 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Functional Gastrointestinal Disorders
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Internet-delivered CBT (Experimental): Children and parents will receive 10 weekly modules of internet-delivered CBT (Cognitive Behavior Therapy). Parents will also receive 10 weekly specific modules for parents. Main components in the modules directed at children and parents are exposure for symptoms, feared stimuli and situations. The parents modules contain information on how they can support their children in the treatment and is based on social learning theory. Therapist support is provided through written messages within the secure platform. Therapists are trained CBT-psychologists.
  Interventions: Behavioral: Internet-delivered CBT

INTERVENTIONS:
Behavioral: Internet-delivered CBT — The treatment is based on an internet-delivered CBT-treatment for adults with IBS and on the adapted version for adolescents with functional gastrointestinal disorders. The protocol has been tested in an open face-to-face CBT study of children aged 8-12 years (n=20) with promising results.
  Main component in the treatment is exposure for symptoms. The purpose of the treatment is to reduce fearful and anxious responses to symptoms and lessen avoidance of symptoms in the child, and to teach the parents how parental behavior can influence symptoms in children as well as how to support exposure. Detailed behaviour analysis is made for each individual and instruction is given on how to gradually expose to symptoms to lessen fear for symptoms and widen the behavioral repertoire.

SUMMARY:
This pilot-study aims to evaluate the effect size and feasibility of internet-delivered cognitive behavior therapy (ICBT) for children (age 8-12 years) with pain-predominant functional gastrointestinal disorders (e.g. irritable bowel syndrome, functional abdominal pain and functional dyspepsia according to the Rome III criteria). The main component investigated in this study is exposure for gastrointestinal symptoms and for feared stimuli and situations. Children will participate along with one of their parents in the treatment. The parents will also receive specific modules with information on how to support their child in the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children between 8-12 years (until their 13th birthday) who have been diagnosed with any of the diagnoses irritable bowel syndrome, functional dyspepsia or functional abdominal pain according to the Rome III criteria.
* Any psychopharmacological medication should be stable since 1 month.
* Parents and children need to master Swedish, have access to a computer with internet access, and be willing to participate in 10 weeks of treatment with homework.

Exclusion Criteria:

* Simultaneous presence of serious somatic disease and / or if the child meets the criteria for other organic disease which better explains the symptoms.
* Psychiatric or social problems that are considered serious and in need of a more intense treatment than ICBT leads to exclusion. Children with higher school absenteeism than 40% will not be included. Neither will children who have an ongoing psychological treatment be included,

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
PedsQL Gastro | Baseline to 10 weeks, baseline to 9 months
  Change in gastrointestinal symptoms measured with a self-rating scale from baseline to 10 weeks, and from baseline to 9 months for analysis of effect.

SECONDARY OUTCOMES:
Faces Pain Rating Scale. (FACES) | Baseline to 10 weeks, baseline to 9 months
  Change in pain intensity measured with a self-rating scale daily during 2 weeks at baseline and daily during 2 weeks after 9 months for analysis of effect.The Faces Pain Scale is a self-report measure used to assess the intensity of children's pain. Faces have four faces representing least pain and most pain on equal intervals on a scale from 0-10. Its validity is supported by a strong positive correlation (r=0.93, N=76) with a visual analogue scale (VAS) measure in children aged 5-12 years. The metric for scoring (0-10) conforms closely to a linear interval scale.
Faces Pain Rating Scale. (FACES) | Weekly during treatment (treatment week 1-9)
  Change in pain intensity measured with a self-rating scale weekly during treatment for mediation analyses.
The Pain App | Baseline to 10 weeks, baseline to 9 months
  Change in pain intensity and daily frequency reported daily during two weeks at baseline, after treatment and at 9 months with a mobile phone application developed by the research group.
Pediatric Quality of Life Inventory (PedsQL) | Baseline to 10 weeks, baseline to 9 months
  Change in quality of life from baseline to 10 weeks, baseline to 9 months measured with a self-report scale that measures quality of life in adolescents. PedsQL Generic Core scales is a 23-item scale ranging from 0 (never) to 4 (almost always). The PedsQL is shown to distinguish between healthy children and adolescents and pediatric patients with acute or chronic health conditions and demonstrate acceptable reliability and validity.
Children´s Somatization Inventory (CSI 24) | Baseline to 10 weeks, baseline to 9 months
  Change in inner symptoms from baseline to 10 weeks, baseline to 9 months, measured with a self-report scale that measures inner symptoms (e.g., headache, nausea, heart racing) that often, but not necessarily, occur in the absence of identified disease, in children and adolescents. CSI-24 is a 24-item scale ranging from ranging from 0 '(not at all) to 4 (a whole lot).
Functional Disability Index (FDI) | Baseline to 10 weeks, baseline to 9 months
  Change in school attendance from baseline to 10 weeks, baseline to 9 months measured with 2 items from a self-report scale that measures school attendance.
Insomnia Severity Index (ISI) | Baseline to 10 weeks, baseline to 9 months
  Change in problematic sleeping patterns from baseline to 10 weeks, baseline to 9 months measured with a self-report scale that measures sleeping habits.
IBS-behavioral responses questionnaire (IBS-BRQ) | Baseline to 10 weeks, baseline to 9 months
  Change in Gastrointestinal symptom-specific behaviors measured with a self-rating scale weekly during treatment for mediation analyses, and from baseline to 10 weeks, baseline to 9 months, for analysis of effect.
Spence Children Anxiety Scale - short version (SCAS) | Baseline to 10 weeks, baseline to 9 months
  Change in anxiety symptoms from baseline to 10 weeks, baseline to 9 months with a self-report scale that measures anxiety symptoms in children and adolescents.
Child Depression Inventory - short version (CDI-S) | Baseline to 10 weeks, baseline to 9 months
  Change in level of depression from baseline to 10 weeks and from baseline to 9 months measured with a self-report scale that measures depression in children and adolescents.
Pain Response Inventory (PRI) - subscale Coping | Baseline to 10 weeks, baseline to 9 months
  Change in pain coping from baseline to 10 weeks and from baseline to 9 months measured with a self-report scale that measures pain coping strategies.
Pressure Activation Stress Scale (PAS) | Baseline to 10 weeks, baseline to 9 months
  Change in stress levels från baseline to 10 weeks and från baseline to 9 months measured with a self-report scale that measures perceived stress. The PAS is developed for children and validated for the age group.
Visceral Sensitivity Index (IBS-VSI) | Baseline to 10 weeks, baseline to 9 months
  Change in visceral sensitivity from baseline to 10 weeks, baseline to 9 months measured with a self-report scale that measures gastrointestinal symptom-specific anxiety.
Client satisfactory questionnaire (CSQ) | At 10 weeks
  Self-rating scale that measures satisfaction with treatment after completion.
Subjective Assessment Questionnaire (SAQ) | At 10 weeks
  Self-rating scale that measures subjective change in symptoms as an effect of treatment.
PedsQL Gastro | Weekly during treatment (treatment week 1-9)
  Change in gastrointestinal symptoms measured with a self-rating scale weekly during treatment for mediation analyses.
IBS-behavioral responses questionnaire (IBS-BRQ) | Weekly during treatment (treatment week 1-9)
  Change in gastrointestinal symptoms-specific behavior measured with a self-rating scale weekly during treatment for mediation analyses.
ROME-III Questionnaire | Baseline to 10 weeks, baseline to 9 months
  Change in children's functional gastrointestinal disorders diagnostic status measured by ROME-III as a self-rating scale.
Adverse Events (AE) | At 10 weeks
  Self-rating scale that measures adverse events related to treatment.
Generalized Anxiety Disorder Screener (GAD-7) | Baseline to 10 weeks, baseline to 9 months
  Change in anxiety levels in parents from baseline to 10 weeks, baseline to 9 months measured with a self-report scale that measures anxiety symptoms. GAD-7 is a 7-item scale ranging from 0 (not at all) to 3 (almost every day). Evidence supports reliability and validity of the GAD-7 as a measure of anxiety in the general population.
Patient Health Questionnaire (PHQ 9) | Baseline to 10 weeks, baseline to 9 months
  Change in depression levels in parents from baseline to 10 weeks, baseline to 9 months measured with a self-report scale that measures depression. PHQ-9 is shown to be a reliable and valid measure of depression severity in adults.
Adult Responses to Children's Symptoms (ARCS) | Baseline to 10 weeks, baseline to 9 months
  Change in parents responses to their children's abdominal pain from baseline to 10 weeks, baseline to 9 months measured with a self-report scale assessing protectiveness, minimizing, and encouraging responses to children's pain behavior.
Parental Behavior in Response to Children's Functional Gastrointestinal Disorders | Baseline to 10 weeks, baseline to 9 months
  Change in parental behavior from baseline to 10 weeks, baseline to 9 months measured with a self-report scale assessing common responses to children´s gastrointestinal symptoms.
Parental Behavior in Response to Children's Functional Gastrointestinal Disorders | Weekly during treatment (treatment week 1-9)
  Change in parental behavior measured weekly with a self-report scale assessing common responses to children´s gastrointestinal symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Ola Olén, MD PhD, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Child and Adolescent Psychiatry in Stockholm, Stockholm, Stockholms Lans Landsting
  - Child and Adolescent Psychiatry in Stockholm, Stockholm